CLINICAL TRIAL: NCT04114045
Title: Effects of Post-exercise Protein Supplementation on Performance Recovery, Muscle Damage, Inflammation and Bone Turnover in Adolescent Swimmers
Brief Title: Effects of Post-exercise Protein Supplementation in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, PKlentrou, Professor and Associate Dean, Brock University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-279 Klentrou
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Fatigue; Inflammation; Bone Resorption
MeSH Terms: conditions — Fatigue; Inflammation; Bone Resorption

STUDY DESIGN:
Intervention Model Description: Participants were divided into three groups: PRO (0.3g/kg - whey protein isolate), CHO (0.3g/kg - maltodextrin) or placebo control (H2O), matched for age, sex and body mass
Who Masked: Participant, Investigator
Masking Description: One member of the research team whom did not have direct contact with participant during performance testing, matched participants for age, sex and body mass into one of three groups (protein, carbohydrate or placebo/water). This member of the research team also prepared and distributed all the research supplements in a sealed black opaque containers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein (Experimental): Whey protein isolate
  Interventions: Dietary Supplement: Experimental:Whey protein
- Isoenergetic control - Carbohydrate (Active Comparator): Carbohydrate or maltodextrin
  Interventions: Dietary Supplement: Active Comparator: Isoenergetic control - Carbohydrate
- Placebo control - Water (Placebo Comparator): Water - chocolate flavoured
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Experimental:Whey protein — Each participant in the protein group received 2 protein drinks immediately following exercise. The supplement was given using a relative quantity of whey protein isolate (0.3g/kg) and was chocolate flavoured.
  Arms: Whey protein
Dietary Supplement: Active Comparator: Isoenergetic control - Carbohydrate — Each participant in the carbohydrate group received 2 drinks immediately following exercise. The supplement was given using a relative quantity of maltodextrin (0.3g/kg), non-caloric chocolate flavouring was added to mask the drinks contents.
  Arms: Isoenergetic control - Carbohydrate
Other: Placebo — Each participant in the water group received 2 drinks immediately following exercise. The water was provided in a similar volume using the same non-caloric chocolate flavouring as the other drinks.
  Arms: Placebo control - Water

SUMMARY:
This randomised double blind, placebo-controlled study examined the effects of post-exercise consumption of whey protein (PRO) or carbohydrate (CHO) on performance recovery, muscle damage and inflammatory cytokine responses following a high intensity interval swim (HIIS) in 10-17-year old male and female swimmers.

DETAILED DESCRIPTION:
Study Procedures: All tests and measurements were performed during three visits at the given swim teams training/practice facility.

During Visit 1, participants were informed of all tests and procedures that will take place and were familiarised with all testing protocols. All anthropometric measurements were also performed during this meeting (see below). Visit one took ~ 60-90 minutes.

During visit 2, Participants arrived at the testing centre for 06:00h, provided a fasted venous blood sample (for biochemical markers - see below). Following the saliva and blood samples, a light breakfast (~300-400 kcal, depending on body mass) (e.g. banana, apple, plain granola bar, water etc.) was provided. Following breakfast (approximately 45-60 min),all participants performed a standardised warm-up in the pool (1000m - short course) followed by 5min of rest and the subsequent performance test in the form of a maximal 200m-front-crawl. Following the maximal 200m performance test, participants underwent a maximal high intensity interval swim protocol (HIIS). The HIIS consisted of 15 high-intensity swimming repetitions (5x100m, 5x50m and 5x25m at maximal intensity) with a work-to-rest ratio of 1:1. Immediately following the HIIS participants exited the pool and provided a second blood sample (blood samples were collected pre-, 30min, 2, 6 and 24h post-HIIS). This was then followed by the first supplement drink ~30-40. 1.5h after consuming the first supplement drink, participants returned to the pool to complete a second maximal 200m swim, followed by a blood test and received their second supplement drink. 1.5h following the supplement drink, a standardised vegetarian lunch was provided, 1.5h following lunch participant provided another blood sample and performed the final 200m swim of that day. Prior to departure participants were provided with a food record sheet to track all food consumption that evening and were instructed to return it to a study investigator the following day.

During visit 3, Participants returned to the testing location at 06:00h, provided a fasted Blood and saliva samples, were given the same breakfast as they received on day 2 and were administered a muscle soreness questionnaire. Following breakfast (approximately 45-60 min),all participants performed the same standardised warm-up as they did in day 2 (1000m - short course) followed by 5min of rest and the subsequent performance test in the form of a maximal 200m-front-crawl.

Groups and supplementation protocol - Participants matched into one of three groups: Protein (0.3g/kg - whey protein isolate), Carbohydrate (0.3g/kg - maltodextrin) or placebo control (flavoured water) (H2O), matched for age, sex and body mass. All groups consumed a total of two supplements, both the investigators and the participants themselves were blinded to the contents of the drink. All drinks were chocolate flavoured and served in black opaque protein shaker cups. For the protein and carbohydrate groups, each participant received an isoenergetic amount of supplement (2 x 0.3g/kg - whey protein isolate or maltodextrin) throughout the duration of the study at the given time-points outlined above.

Biochemical measurements:

Venous blood samples and a saliva sample will be collected on 5 separate occasions (pre-, 30min, 2, 6 and 24h post-HIIS). To control for circadian rhythm, the exercise session and related blood samples will be performed at the same time of day.

Venous blood samples were collected from the antecubital fossa of each participant using a standard venipuncture technique. Endocrine response such as anabolic/hormonal markers, inflammatory markers (cytokines - IL-6, IL-10, TNF-α) and indicators of muscle fatigue/damage (CK) were examined.

ELIGIBILITY:
Inclusion Criteria:

* competitive swimmers (swim competitively for a minimum of 2y)
* male or female 11-17y
* free from any medical conditions

Exclusion Criteria:

* yes on medical screening questionnaire
* not classified as a competitive swimmer (swim competitively for <2y)
* outside the desired age range (<11 or >17)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Performance recovery | 24 hours
  200m front crawl time (s) measured in short course pool (25m)
IL-6 (pg/ml) | 24 hours
  Myokine
IL-10 (pg/ml) | 24 hours
  Anti-inflammatory cytokine
TNF-alpha (pg/ml) | 24 hours
  Pro-inflammatory cytokines
Muscle damage | 24 hours
  Creatine kinase activity (u/L)
Bone formation marker | 24 hours
  Procollagen type 1 intact N-terminal propeptide, PINP (ng/ml)
Bone resorption marker | 24 hours
  Carboxy-terminal collagen crosslinks, CTXI (ng/ml)

SECONDARY OUTCOMES:
Bone turnover balance | 24 hours
  Balance between bone formation and resorption calculated from the ratio of Median (PINP)/Median(CTXI)
Rate of Bone turnover | 24 hours
  Rate of bone formation and resorption calculated as √[MoMF(square) + MoMR(square)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Klentrou, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, Saint Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McKinlay BJ, Theocharidis A, Adebero T, Kurgan N, Fajardo VA, Roy BD, Josse AR, M Logan-Sprenger H, Falk B, Klentrou P. Effects of Post-Exercise Whey Protein Consumption on Recovery Indices in Adolescent Swimmers. Int J Environ Res Public Health. 2020 Oct 23;17(21):7761. doi: 10.3390/ijerph17217761. PMID 33114186
- [Result] Theocharidis A, McKinlay BJ, Vlachopoulos D, Josse AR, Falk B, Klentrou P. Effects of post exercise protein supplementation on markers of bone turnover in adolescent swimmers. J Int Soc Sports Nutr. 2020 Apr 15;17(1):20. doi: 10.1186/s12970-020-00350-z. PMID 32293471
- [Result] Sanderson M, McKinlay BJ, Theocharidis A, Kouvelioti R, Falk B, Klentrou P. Changes in Inflammatory Cytokines and Irisin in Response to High Intensity Swimming in Adolescent versus Adult Male Swimmers. Sports (Basel). 2020 Dec 1;8(12):157. doi: 10.3390/sports8120157. PMID 33271764